CLINICAL TRIAL: NCT03452995
Title: Manual Lymphatic Drainage Integrated With Kinesio Tape and Traditional Rehabilitation Techniques in Patients Operated for Knee Arthroplasty in Osteoarthritis
Brief Title: Lymphodreinage Integrated With Kinesio Tape in TKA Patients
Acronym: LINFOTAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Laura Tornatore, Physical Therapist, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0009494
Record Dates: First submitted 2018-02-20; First posted 2018-03-02 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: TOTAL KNEE ARTHROPLASTY; Edema Secondary; Pain; Joint Dysfunction
MeSH Terms: conditions — Pain; Joint Diseases | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physiotherapy: LYMPHO DRAINAGE (Active Comparator): Patients will be treated on the second postoperative day, on the 4th postoperative day and on the 6th post-operative day by means of Manual lymphodrainage consisting in special massage technique that allows lymphatic drainage, or removal of interstitial fluid stagnation according to Vodder, in association to the standard rehabilitation protocol for TKA (Kinetec, functional rehabilitation and walking training
  Interventions: Procedure: PHYSIOTHERAPY
- Physiotherapy: KINESIOTAPING (Active Comparator): Patients will be treated on the second postoperative day, on the 4th postoperative day and on the 6th post-operative day through the use of patches acting through the sensory system giving stimuli to receptors on the skin, in association to the standard rehabilitation protocol for TKA (kinetec, functional rehabilitation and walking training .
  Interventions: Procedure: PHYSIOTHERAPY
- Physiotherapy:LYMPHO+KINESIO (Experimental): Patients will ne treated with both kinesiotaping and lymphodreinage on the second post-operative day, on 4 days post-operative and on the 6th post-operative day, in association to the standard rehabilitation protocol for TKA (kinetec, functional rehabilitation and walking training
  Interventions: Procedure: PHYSIOTHERAPY

INTERVENTIONS:
Procedure: PHYSIOTHERAPY — Lymphodreinage and kinesiotaping are current methods of treatment of edema, pain and indirectly recovery of the knee ROM in TKA. Edema, pain and knee ROM are strictly corelated and, by reducing edema, we reduce the pressure by relieving pain, and allowing an improvement in movement.
  Other Names: Lymphodreinage, kinesiotaping

SUMMARY:
Aim of the study: To evaluate the efficacy of lymphatic drainage treatment associated with the application of kinesiotaping in the reduction of lymphedema, pain and in the recovery of knee joint ROM in patients undergoing surgery of total knee arthroplasty in osteoarthritis.

Inclusion criteria: Operated patients of total primary knee arthroplasty in osteoarthritis not later than 5 days after surgery, Patients of both sexes aged between 65 and 85, Presence of lymphedema and volumetric difference with the contralateral limb of the cirtometry equal or greater than 3 cm.

Exclusion criteria: Patients operated for re-implantation or revision, presence of inflammatory, neurological, important cardiological diseases and active tumor pathologies, absence of DVT of the lower limb.

Study design: Prospective, open, randomized, lasting 12 months GROUP 1 (33 pts) KINESIOTAPING + STANDARD REHABILITATION GROUP 2 (33 pts) LYMPHODRAINAGE+ STANDARD REHABILITATION GROUP 3 (33 pts) KINESIOTAPING + LYMPHODRAINAGE + STANDARD REHABILITATION Outcome measures: Pain: evaluation with NRS scale 0-10, Edema: cirtometric evaluation (in 4 standard points), ROM: goniometric measurement of the knee joint excursion. All measures at the beginning and end of treatment (6 days).

DETAILED DESCRIPTION:
Background In the days following knee arthroplasty, the presence of a strong local inflammatory component is associated with pain and functional limitation, which usually resolves within a few months; however, sometimes it can take longer, and sometimes result in a condition of chronic inflammation, albeit modest, that lasts for years. Lymphodrainage and Kinesiotaping have been indicated as effective treatments to reduce edema and alleviate pain. However it is not clear which of these techniques is more effective and if their effectiveness increases when combined.

Objective of the study The objective of the study is to evaluate the effectiveness of lymphatic drainage treatment associated with the application of kinesiotaping in the reduction of lymphedema, pain and in the recovery of knee joint excursion (ROM) in patients undergoing total arthroplasty knee in osteoarthritis. The hypothesis is that the associated treatment of kinesiotaping and lymphatic drainage produces better results than the individual treatments.

Methods

Patients will be divided in 3 groups according to the type of treatment:

GROUP 1 Lymphatic drainage + standard rehabilitation GROUP 2 Kinesiotaping + standard rehabilitation GROUP 3 Lymphatic drainage + Kinesiotaping + standard rehabilitation For each patient the duration of the study will be 6 days, the total duration of the study will be 12 months.

Statistics Considering the NRS for the evaluation of pain as a primary outcome, the determination of the sample was made on the basis of the following assumptions: level of significance (α) = 0.05, (2) type 2 error (β) = 0.2; with an 80% test power ,.

For the calculation of the sample G * Power 3.1.7 was used based on an effect size of 0.8 (Large effect size according to Cohen) and the Bonferroni correction for multiple comparisons. The calculated dimension of the sample was thus determined of 30 patients per group. Considering a drop-out of 10% the total sample should be 99 patients (33 per group). All continuous variables will be expressed in terms of mean ± standard deviation (SD) and range. To analyze the data collected, one-way analysis will be used with a post hoc comparison test for paired Sidak data. Statistical analysis will be performed with SAS / Stat software (version 9.3; SAS Institute, Cary, North Carolina). For all tests a P <0.05 will be considered significant.

Treatment All enrolled patients will receive a standard rehabilitation treatment consisting of

* KINETEC 1 h / day
* Functional rehabilitation 30 min for 2 times/day
* Walking training 15 min for 2 times/day

For each of the three groups experimental treatments will be added

GROUP 1 Lymphodrainage + elastic containment (postoperative compression stockings), 3 treatments: in the second postoperative day, in 4th postoperative day and in 6th post-operative day

GROUP 2 Kinesiotaping, 3 treatments: in the second postoperative day, in 4th postoperative day and in 6th post-operative day

GROUP 3 Lymphodrainage and Kinesiotaping, 3 treatments: on the second post-operative day, on 4 days post-operative and on the 6th post-operative day

The Vodder massage technique will be used for lymphatic drainage. The peculiarity of this method is the absolute respect of the lymphatic directions, of the operative pressures, of the frequency, of the rhythm and of the gesture. The various manoevers on the different body districts are performed in a proximal-distal sense, to respect the lymphatic course in directions of the lymph node stations and are performed with harmonic, slow and rhythmic movements. Manual pressures should not exceed 30-40 mmHg, but may vary depending on the consistency of the edema. In the specific case of the project, drainage is followed in the lower limb of the anterior and posterior part by placing the neck ganglia empty, which is peculiar to the original Volder method, used for about 30 minutes.

As for the Kinesiotaping as a lymphatic application the fan technique applied in the back of the thigh and the leg, and in the front of the foot (back of the foot) will be used with the aim of activating the cutaneous mechanoreceptors, reduce the pressure at the level interstitial in order to promote lymphatic drainage and ensure that this application leads to the reduction of swelling of post-operative soft tissues.

Adverse events The expected techniques do not foresee adverse events therefore, considering the good tolerance of the patients and the scarcity of known contraindications, we can state that the treatment is safe and can be an additional measure for pain reduction as well as edema. However, it is possible that the areas treated with neuromuscular tape may show skin irritations caused by the glue of the tape in case of very delicate skin.

ELIGIBILITY:
Inclusion Criteria:

* Operated patients of total primary knee arthroplasty in osteoarthritis not later than 5 days after surgery
* Patients of both sexes aged between 65 and 85;
* Presence of lymphedema and volumetric difference with the contralateral limb of the cirtometry equal or greater than 3cm.

Exclusion Criteria:

* Patients operated for re-implantation or revision
* Presence of inflammatory, neurological, important cardiological diseases and active tumor pathologies.
* Absence of DVT of the lower limb.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Pain severity | Change between baseline and the end of treatment (6 days)
  NRS Pain: the Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain.
  Pain Level rating:
  0 No Pain 1-3 Mild Pain 4-6 Moderate Pain 7-10 Severe Pain

SECONDARY OUTCOMES:
Edema | Change between baseline and the end of treatment (6 days)
  cirtometric evaluation (in 3 standard points (above the knee: 10 cm above the upper patellar pole, 10 cm below the inferior patellar pole, ankle).
KNEE ROM | Change between baseline and the end of treatment (6 days)
  goniometric measurement of the knee joint excursion operated at the beginning and end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laura Tornatore, PT, Principal Investigator — Istituto Ortopedico Rizzoli DRS
Locations (1):
- Istituto Ortopedico Rizzoli DRS, Bagheria, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No